CLINICAL TRIAL: NCT04383951
Title: Safety and Efficacy of Ketogenic Diet for Promoting Weight Loss in Obese Individuals With Compensated NASH Cirrhosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Raj Vuppalanchi, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Keto Diet Study
Record Dates: First submitted 2020-04-17; First posted 2020-05-12 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; Cirrhosis, Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Block randomization will be utilized to ensure balancing of treatment groups throughout enrollment. 30 participants will be assigned to the ketogenic diet arm and 10 will be assigned to standard of care.
Who Masked: Investigator
Masking Description: While this is an open label study, the principal investigator will be blinded to the results of efficacy outcomes such as MRI-PDFF, Body composition data, VCTE by FibroScan® and study questionnaires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet (Active Comparator): For participants randomized to the ketogenic diet arm, a consultation with the providers of medically supervised weight loss clinic of Indiana University Health will be arranged. Subjects will be educated on the concepts of ketosis, symptoms associated with it, and dietary manipulation to achieve ketosis. Participants in this arm will use the suggested recipes in combination with strict carbohydrate monitoring though checking for urine ketone bodies. These recipes were gathered and vetted by the dietitian at the medically supervised weight loss clinic. We anticipate that this approach will allow for more calorie intake and easier carbohydrate restriction. The follow up visits will be determined by the providers of the medically supervised weight loss clinic based on the symptoms reported and subject's compliance with carbohydrate restriction.
  Interventions: Other: Dietary consult for participants in the ketogenic diet arm
- Standard of Care (Sham Comparator): For participants randomized to this arm, a consultation with the providers of medically supervised weight loss clinic will be arranged. The discussion will focus on portion control using a balanced diet. A follow up visit will be at 16 weeks. This is the extent of interventions received for participants in this arm.
  Interventions: Other: Dietary consult for participants in the standard of care arm

INTERVENTIONS:
Other: Dietary consult for participants in the ketogenic diet arm — An initial consultation with the providers of medically supervised weight loss clinic will be arranged. Participants in the ketogenic diet group will be educated on the concepts of the diet and will be provided with recipes to be utilized at home that adhere to this diet. In addition to the initial consultation, participants in this arm receive additional consultations with these providers with a frequency as determined by the provider.
  Arms: Ketogenic diet
Other: Dietary consult for participants in the standard of care arm — For participants in the standard of care arm, an initial consultation with the providers of medically supervised weight loss clinic will be arranged and the discussion will center around portion control using a balanced diet. Participants will receive only one additional consultation with the provider 16 weeks later just prior to the conclusion of the study.
  Arms: Standard of Care

SUMMARY:
This is an open-label, randomized study comparing a monitored ketogenic diet intervention using standard ketogenic diet (SKD) and standard of care (SOC) dietary recommendations for 16 weeks. Subjects enrolled in the standard of care group will receive a voucher to Weight Watchers after study completion.

DETAILED DESCRIPTION:
The primary aim is to assess the safety of ketogenic diet as compared to standard of care approach for weight loss in patients with compensated cirrhosis due to NASH. The safety endpoints captured in the study include liver decompensation events, measured through several questionnaires, fasting blood glucose, serum creatinine, fasting lipid profile and other adverse events. The tolerability of the ketogenic diet will be assessed by study compliance and by administering a questionnaire.

Secondary aims include weight loss, changes in body composition via serial use of bioelectrical impedance via an Inbody Machine, changes in liver fat and liver stiffness using MRI and proton density fat fraction (MRI-PDFF), liver biochemistries, changes in Child-Turcotte-Pugh and MELD scores measured via labs and changes in liver steatosis and stiffness via serial measures of VCTE by FibroScan®.

ELIGIBILITY:
Inclusion Criteria:

1. NASH cirrhosis (criteria in Appendix 1) with obesity (BMI >30 kg/m2).
2. Age 18 and greater

Exclusion Criteria:

1. Actively participation in investigational drug treatment for non-alcoholic fatty liver disease
2. Currently taking medications for weight loss or have joined a supervised weight loss program prior to enrollment
3. Have hepatocellular carcinoma and are undergoing therapy
4. Women who become pregnant or plan to become pregnant prior to the study date; female subjects who become pregnant during the study will be withdrawn from the study
5. Pacemaker or implantable cardioverter devices
6. History of hepatic surgery
7. Current significant alcohol consumption, defined as more than 20 grams per day in females or 30 grams per day in males
8. Presence of ascites or hepatic encephalopathy
9. Symptomatic gastroparesis
10. Uncontrolled diabetes, as defined by a HgbA1C >11%
11. Uncontrolled congestive heart failure
12. Active infections
13. Child Turcotte Pugh score > 6
14. MELD score >12
15. Unwilling to undergo an MRI or have contraindications to an MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood chemistry to assess for liver de-compensation events | Blood chemistry tests will be assessed at the initial visit.
  Blood will be drawn serially to assess fasting blood glucose, serum creatinine and fasting lipid profile.
Blood chemistry to assess for liver de-compensation events | Blood chemistry tests will be assessed at the study visits between weeks 5 and 14.
  Blood will be drawn serially to assess fasting blood glucose, serum creatinine and fasting lipid profile.
Blood chemistry to assess for liver de-compensation events | Blood chemistry tests will be assessed at the Week 16 visit.
  Blood will be drawn serially to assess fasting blood glucose, serum creatinine and fasting lipid profile.
Adverse events | All participants will be monitored at the study visits between weeks 5 and 14 and all participants will be instructed to alert the study team for additional information if such an event occurs.
  All participants will be monitored for adverse events and/or serious adverse events throughout the duration of the trial.
Adverse events | All participants will be monitored at the week 16 visit and all participants will be instructed to alert the study team for additional information if such an event occurs.
  All participants will be monitored for adverse events and/or serious adverse events throughout the duration of the trial.
Tolerability of the ketogenic diet | The POMS 40 questionnaire is administered at the initial visit.
  How well the ketogenic diets is tolerated will be assessed by administering a POMS40 questionnaire.
Tolerability of the ketogenic diet | The POMS 40 questionnaire is administered at the study visits between weeks 1 and 4.
  How well the ketogenic diets is tolerated will be assessed by administering a POMS40 questionnaire.
Tolerability of the ketogenic diet | The POMS 40 questionnaire is administered at the Week 16 visit.
  How well the ketogenic diets is tolerated will be assessed by administering a POMS40 questionnaire.

SECONDARY OUTCOMES:
MRI with proton density fat fraction (PDFF) | Performed at initial visit and at week 16 visit
  MRI-PDFF is a convenient method for liver fat quantification and currently used in most clinical trials, as it only requires a single 20-second breath hold and an estimated time of about 5 minutes in an MRI scanner suite. MRI in the study will be used to quantify liver steatosis, stiffness, and body composition.
Weight loss and change in body composition | Performed at initial visit and at week 16 visit
  Changes in weight and body composition will be measured via serial use of a scale and use of bioelectrical impedance via an Inbody machine
Changes in liver stiffness and steatosis | Performed at initial visit and at week 16 visit
  Changes in liver stiffness and steatosis will be measured with serial use of vibration controlled transient elastography (VCTE) via a FibroScan.

CONTACTS AND LOCATIONS:
Overall Officials: Raj Vuppalanchi, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No IPD at this time